CLINICAL TRIAL: NCT02581124
Title: A Phase 1, Open-label Study to Evaluate the Effect of Lapatinib, a BCRP Inhibitor, on the Pharmacokinetics of JTZ-951 in Subjects With End-stage Renal Disease Receiving Hemodialysis
Brief Title: Study to Evaluate Effect of Lapatinib on Pharmacokinetics of JTZ-951 in Subjects With End-stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ951-U-15-009
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: JTZ-951; Lapatinib; Pharmacokinetics
MeSH Terms: interventions — enarodustat; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: JTZ-951 and Lapatinib (Experimental): Tablets; JTZ-951, single dose on non-dialysis Days 1 and 5; Lapatinib, single dose on non-dialysis Day 5
  Interventions: Drug: JTZ-951; Drug: Lapatinib

INTERVENTIONS:
Drug: JTZ-951
Drug: Lapatinib

SUMMARY:
Study to evaluate the effect of lapatinib, a breast cancer resistance protein (BCRP) inhibitor, on the pharmacokinetics (PK) of JTZ-951 and to evaluate the safety and tolerability of JTZ-951 when administered alone and one hour after the administration of lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end stage renal disease on hemodialysis
* Post-dialysis body weight >45.0 kg
* BMI between 18.0 and 40.0 kg/m2 (inclusive)

Exclusion Criteria:

* Subjects with positive test results for HBsAg (hepatitis B surface antigen), HCV antibody or HIV antibody
* Subjects with known history of liver failure or liver surgery
* Subjects with a history or current clinically significant chronic or acute blood loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration) | 10 days
tmax (time to reach maximum concentration) | 10 days
AUC (area under the concentration-time curve) | 10 days
t1/2 (elimination half-life) | 10 days
Number of adverse events | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis, Minnesota, United States